CLINICAL TRIAL: NCT01597895
Title: Open-Label, Randomized, Fixed-Sequence, Crossover Study to Estimate the Effect of Telaprevir and Boceprevir on Maraviroc Pharmacokinetics in Healthy Subjects
Brief Title: Estimate the Effect of Telaprevir and Boceprevir on Maraviroc Pharmacokinetics in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A4001108
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: maraviroc; boceprevir; telaprevir; drug interaction; pharmacokinetics; HIV
MeSH Terms: interventions — Maraviroc; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Maraviroc (Active Comparator)
  Interventions: Drug: Maraviroc
- Maraviroc + Boceprevir (Experimental)
  Interventions: Drug: Maraviroc + Boceprevir
- Maraviroc + Telaprevir (Experimental)
  Interventions: Drug: Maraviroc + Telaprevir

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 150 mg BID x 5 days with food
  Arms: Maraviroc
Drug: Maraviroc + Boceprevir — Maraviroc 150 mg BID + Boceprevir 800 mg TID x 10 days with food
  Arms: Maraviroc + Boceprevir
Drug: Maraviroc + Telaprevir — Maraviroc 150 mg BID + Telaprevir 800 mg TID x 10 days with food
  Arms: Maraviroc + Telaprevir

SUMMARY:
The purpose of this study is to determine the effect that telaprevir and boceprevir has on the pharmacokinetics of maraviroc.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.
* Total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Positive result for HIV-1, HIV-2, Hepatitis B serology (HbsAg, HbcAb) or anti hepatitis C virus serology (as determined by a multi antigen EIA).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maraviroc plasma pharmacokinetic parameters: AUC12, Cmax, and C12h on Period 1, Day 5 and Periods 2 and 3, Day 10 | 25 days

SECONDARY OUTCOMES:
Maraviroc plasma pharmacokinetic parameters: Tmax on Period 1, Day 5 and Periods 2 and 3, Day 10 | 25 days
Boceprevir plasma pharmacokinetic parameters: AUC8, Cmax, C8h, and Tmax on Period 2, Day 10 | 10 days
Telaprevir plasma pharmacokinetic parameters: AUC8, Cmax, C8h, and Tmax on Period 3, Day 10 | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001108&StudyName=Estimate%20the%20Effect%20of%20Telaprevir%20and%20Boceprevir%20on%20Maraviroc%20Pharmacokinetics%20in%20Healthy%20Subjects%20